CLINICAL TRIAL: NCT01534546
Title: A Randomized, Multicenter, Controlled Phase III Study to Compare Perioperative Chemotherapy of Oxaliplatin Combined With S-1(SOX) Versus SOX or Oxaliplatin With Capecitabine (XELOX) as Post-operative Chemotherapy in Locally Advanced Gastric Adenocarcinoma With D2 Dissection
Brief Title: Phase III Study to Compare Perioperative Chemotherapy of Oxaliplatin Combined With S-1(SOX) Versus SOX or Oxaliplatin With Capecitabine (XELOX) as Post-operative Chemotherapy in Locally Advanced Gastric Adenocarcinoma With D2 Dissection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, head of Department of gastrointestinal oncology, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG1003-RESOLVE; CGOG 1003 (Other: Chinese Gastrointestinal Oncology Group)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Advanced Gastric Carcinoma
Keywords: neoadjuvant chemotherapy; adjuvant chemotherapy; DFS; OS; safety; resectable locally advanced gastric carcinoma; potentially resectable locally advanced gastric carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- arm A postoperative Oxaliplatin/capecitabine（XELOX） (Active Comparator): postoperative Oxaliplatin/capecitabine（XELOX） patients in arm A will receive standard gastrectomy with D2 Lymphadenectomy first, and 8 cycles of adjuvant XELOX later.
  capecitabine：1000 mg/m2 ，bid, d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W 8 cycles (6 months)
  Interventions: Drug: Oxaliplatin capecitabine
- arm B: postoperative Oxaliplatin/S-1（SOX） (Experimental): postoperative Oxaliplatin/S-1（SOX） patients in arm B will receive standard gastrectomy with D2 Lymphadenectomy first, and 8 cycles of adjuvant SOX later.
  S-1：40~60mg bid，d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W 8 cycles (6 months)
  Interventions: Drug: Oxaliplatin S-1
- Arm C：postoperative Oxaliplatin /S-1（SOX） (Experimental): Postoperative Oxaliplatin /S-1（SOX） patients in arm C will receive 3 cycles of neoadjuvant SOX first, and then standard gastrectomy with D2 lymphadenectomy, and 5 cycles of adjuvant SOX followed by 3 cycles of S-1 monotherapy.
  Dose of s-1 and oxaliplatin are same to arm B Dose of S-1 monotherapy is same to combination therapy (SOX 3 cycles before surgery, 5 cycles of SOX and 3 cycles of S-1 monotherapy, 6 months after surgery)
  Interventions: Drug: Oxaliplatin S-1

INTERVENTIONS:
Drug: Oxaliplatin capecitabine — capecitabine：1000 mg/m2 ，bid, d1~14 oxaliplatin：130mg/m2，iv drip for 2h，d1
  Arms: arm A postoperative Oxaliplatin/capecitabine（XELOX）
Drug: Oxaliplatin S-1 — S-1: 40~60mg bid，po, d1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid） oxaliplatin：130mg/m2，iv drip for 2h，d1
  Arms: arm B: postoperative Oxaliplatin/S-1（SOX）
Drug: Oxaliplatin S-1 — S-1: 40~60mg bid，d1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid） oxaliplatin：130mg/m2，iv drip for 2h，d1 S-1 monotherapy as the same dose and schedule of the above
  Arms: Arm C：postoperative Oxaliplatin /S-1（SOX）

SUMMARY:
Peri-operative treatment of locally advanced gastric cancer (LAGC) has always been argued by eastern and western scholars. For patients with clinical stage of cT4b/N+M0, or cT4aN+M0, the prognosis is rather poor, and the primary lesions might not be resectable at the time of diagnosis. MAGIC study has showed that pre-and post-operative chemotherapy with 3 cycles of ECF has increased 13% on 5yOS compared with surgery alone; However, eastern studies such as ACTS GC or CLASSIC showed that TS-1 monotherapy or XELOX (oxaliplatin/capecitabine) combination given as adjuvant chemotherapy for stage II or III patients after D2 surgery could achieve the significant survival benefit. So whether perioperative or post operative therapy is more beneficial for LAGC patients lacks of data supported by prospective study.

So in this prospective randomized phase III study, the investigators aim to compare the survival benefit as well as the safety for SOX (oxaliplatin/TS-1) as perioperative therapy versus SOX or XELOX as postoperative therapy after D2 dissection.

DETAILED DESCRIPTION:
detailed discription of protocol updated on Feb 2013; detailed discription of protocol updated on Apr 2013; detailed discription of protocol updated on Oct 2013;

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent form
* age ≥ 18 years
* pathologically confirmed gastric or GEJ adenocarcinoma
* disease at clinical stage of resectable or potentially resectable LAGC（T4a-b/N+M0）
* No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
* Adequate organ function as defined below:

Hematologic ANC ≥ 1.5*109/l Hemoglobin ≥ 9 g/dl Platelets ≥ 100*109/l Hepatic Albumin ≥ 30g/l Serum bilirubin ≤ 1.5×ULN AST and ALT ≤ 2.5×ULN ALP ≤ 2.5×ULN TBIL ≤ 1.5×ULN Renal Serum Creatinine < 1.5 ULN

* KPS ≥ 70
* Adequate lung and heart function
* Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women
* Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

* Refuse to provide blood/tissue sample；
* With distant metastasis；
* Sexually active males or females refuse to practice contraception during the study until 30 days after end of study.
* Known hypersensitivity reaction or metabolic disorder to fluorpyrimidines or oxaliplatin；
* ≥ grade 1 peripheral neuropathy；
* History of organ transplantation（including autologous bone marrow transplantation and Peripheral stem cell transplantation）；
* Prior long term steroid therapy (excluding short term steroid treatment which is completed prior to > 2 weeks of study enrollment)；
* Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease；
* Concurrent severe infection；
* unable to swallow; (complete or incomplete)gastrointestinal obstruction; gastrointestinal bleeding; gastrointestinal perforation；
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety (including current active hepatic, biliary, renal, respiratory disease, uncontrolled diabetes hypertension et al)；
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible；
* Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency；
* Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 2012-03; Primary Completion 2019-07 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
3 year Disease Free Survival | 3 years
  1. perioperative chemotherapy of SOX is superior than postoperative SOX after D2 dissection in LAGC.
  2. Postoperative SOX is non inferior to XELOX.

SECONDARY OUTCOMES:
5 year Overall Survival | 5 years
  1. perioperative chemotherapy of SOX is superior than postoperative SOX after D2 dissection in LAGC.
  2. Postoperative SOX is non inferior to XELOX.
Adverse Event | 1year
  peri-operation morbidity, mortality, and other adverse events including chemotherapy related ones.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Lin Shen, Beijing
  - Peking Unicersity Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Liang H, Li Z, Xue Y, Wang Y, Zhou Z, Yu J, Bu Z, Chen L, Du Y, Wang X, Wu A, Li G, Su X, Xiao G, Cui M, Wu D, Chen L, Wu X, Zhou Y, Zhang L, Dang C, He Y, Zhang Z, Sun Y, Li Y, Chen H, Bai Y, Wang Y, Yu P, Zhu G, Suo J, Jia B, Li L, Huang C, Li F, Ye Y, Xu H, Wang X, Yuan Y, E J, Ying X, Yao C, Shen L, Ji J. Perioperative or postoperative adjuvant oxaliplatin with S-1 versus adjuvant oxaliplatin with capecitabine in patients with locally advanced gastric or gastro-oesophageal junction adenocarcinoma undergoing D2 gastrectomy (RESOLVE): final report of a randomised, open-label, phase 3 trial. Lancet Oncol. 2025 Mar;26(3):312-319. doi: 10.1016/S1470-2045(24)00676-4. Epub 2025 Feb 11. PMID 39952264
- [Derived] Zhang X, Liang H, Li Z, Xue Y, Wang Y, Zhou Z, Yu J, Bu Z, Chen L, Du Y, Wang X, Wu A, Li G, Su X, Xiao G, Cui M, Wu D, Chen L, Wu X, Zhou Y, Zhang L, Dang C, He Y, Zhang Z, Sun Y, Li Y, Chen H, Bai Y, Qi C, Yu P, Zhu G, Suo J, Jia B, Li L, Huang C, Li F, Ye Y, Xu H, Wang X, Yuan Y, E JY, Ying X, Yao C, Shen L, Ji J; RESOLVE study group. Perioperative or postoperative adjuvant oxaliplatin with S-1 versus adjuvant oxaliplatin with capecitabine in patients with locally advanced gastric or gastro-oesophageal junction adenocarcinoma undergoing D2 gastrectomy (RESOLVE): an open-label, superiority and non-inferiority, phase 3 randomised controlled trial. Lancet Oncol. 2021 Aug;22(8):1081-1092. doi: 10.1016/S1470-2045(21)00297-7. Epub 2021 Jul 9. PMID 34252374